CLINICAL TRIAL: NCT03783754
Title: Triple Therapy Prevention of Recurrent Intracerebral Disease EveNts Trial (TRIDENT) MRI Sub-study
Brief Title: Triple Therapy Prevention of Recurrent Intracerebral Disease EveNts Trial Magnetic Resonance Imaging Sub-study
Acronym: TRIDENT-MRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not feasible to continue
Sponsor: The George Institute (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: TRIDENT MRI
Record Dates: First submitted 2018-12-06; First posted 2018-12-21 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Stroke; Cerebral Small Vessel Diseases; Intracerebral Hemorrhage; Vascular Dementia; Hypertension
MeSH Terms: conditions — Stroke; Cerebral Small Vessel Diseases; Cerebral Hemorrhage; Dementia, Vascular; Hypertension | interventions — Telmisartan; Amlodipine; Indapamide

STUDY DESIGN:
Intervention Model Description: Main Study: Multicentre, international, double-blinded, placebo-controlled, parallel-group, randomised controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple Pill (Active Treatment) (Experimental): telmisartan 20mg, amlodipine 2.5mg, and indapamide 1.25mg;
  Interventions: Drug: telmisartan 20 mg + amlodipine 2.5mg + indapamide 1.25mg
- Placebo (Placebo Comparator): received via blinded study oral capsules
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: telmisartan 20 mg + amlodipine 2.5mg + indapamide 1.25mg — low-dose combination therapy
  Other Names: Triple Pill
  Arms: Triple Pill (Active Treatment)
Drug: Placebo oral capsule — matched placebo
  Arms: Placebo

SUMMARY:
TRIDENT Main Study:

TRIDENT is a multicentre, international, double-blinded, placebo-controlled, parallel-group, randomised controlled trial of a fixed low-dose combination BP-lowering pill ("Triple Pill") strategy on top of standard of care, in patients with a history of acute intracerebral haemorrhage (ICH) and systolic blood pressure (SBP) levels defined as 'high normal to borderline high', and on either minimal or no BP-lowering treatment according to current guidelines.

MRI Sub-Study Centres capable of specific MRI of the brain sequences will be identified. The patients in the TRIDENT main study who are identified to be eligible for the MRI Sub-Study will undergo MRI scans at baseline (6 weeks to 6 months post-randomisation) and at 36-month follow-up time points. All data collected will be analysed centrally at the Brain and Mind Centre (BMC) in Sydney, Australia.

DETAILED DESCRIPTION:
Intracerebral haemorrhage (ICH) is the most serious type of stroke, accounting for 10% of stroke in high-income countries and up to 50% in low-to-middle income countries, especially in Asia where hypertension is common. ICH in the context of hypertension is often a manifestation of underlying cerebral small vessel disease (CSVD).

In summary, there is a considerable body of evidence supporting and association of CSVD with hypertension and poor outcomes, but limited evidence as to whether good BP control can modify the natural history of this condition.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for, randomised and continuing in TRIDENT Main Study
2. No contraindications to MRI scan of the brain
3. Provide informed consent for the MRI Sub-Study

Exclusion Criteria:

1. Any MRI contraindications (e.g. metallic implants, claustrophobia, etc.)
2. Less than 6 weeks or greater than 6 months post-randomisation (however, where possible the baseline MRI Sub-Study scan should be conducted as soon as possible after the qualifying ICH. e.g. if the qualifying ICH was 4 months prior to randomisation, the baseline scan should be done as close to 6 weeks post-randomisation as possible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-03-21 (Actual)

PRIMARY OUTCOMES:
Change in T2 FLAIR white matter hyperintensities (WMH) volume | 36 months

SECONDARY OUTCOMES:
Whole brain atrophy measured by percentage brain volume change between baseline and 36 months on HIRES-T1. | 36 months
Substructure change - cortical grey matter | 36 months
  expected range: >400,000 and <800,000mm3 Relevant Sequence: 3D-T1
Substructure change - white matter | 36 months
  expected range: >400,000 and <900,000mm3 Relevant Sequence: 3D-T1
Substructure change - cerebrospinal fluid (CSF) | 36 months
  volume change measured Relevant Sequence: 3D-T1
Change in number of cerebral microbleeds (CMBs) | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Craig Anderson, Prof, Principal Investigator — The George Institute
Locations (3):
- Australia (3):
  - Liverpool Hospital, Liverpool, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Melbourne Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No